CLINICAL TRIAL: NCT02051946
Title: Novel Drug Delivery Technique for Glaucoma Patients
Brief Title: Novel Drug Delivery Technique Via Retroject Device
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Molly Walsh (Other)
Responsible Party: Sponsor-Investigator, Molly Walsh, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00039988
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Glaucoma
Keywords: novel drug delivery technique for glaucoma patients
MeSH Terms: conditions — Glaucoma | interventions — Ethacrynic Acid; Hanks Balanced Salt Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Retroject device only (Active Comparator): The first 5 patients enrolled will serve as controls and will have the device alone placed on the eye (without an injection of ethacrynic acid).
  Interventions: Device: Retroject Device
- Retroject injection with ethacrynic acid injection (Experimental): The next 3 patients, after the first 5 controls, will have the device placed on the eye with a subsequent injection of ethacrynic acid into the episcleral vein.
  Interventions: Device: Retroject Device; Drug: ethacrynic acid injection
- randomization to ethacrynic acid or balanced salt solution (Experimental): The last 12 patients will all have the device placed on their eye. They will then be randomized in a 2:1 ratio to receive either an injection of ethacrynic acid or balanced salt solution.
  Interventions: Device: Retroject Device; Drug: ethacrynic acid injection; Drug: balanced salt solution

INTERVENTIONS:
Device: Retroject Device
Drug: ethacrynic acid injection
  Arms: Retroject injection with ethacrynic acid injection; randomization to ethacrynic acid or balanced salt solution
Drug: balanced salt solution
  Arms: randomization to ethacrynic acid or balanced salt solution

SUMMARY:
The purpose of this study is to identify whether or not injection of a study drug (ethacrynic acid) using the investigational Retroject device is able to lower eye pressures in patients with advanced glaucoma. 20 patients with advanced glaucoma with visual acuity less than 20/200 and intraocular pressures (IOP) >20mmHg on maximum medical therapy will be asked to participate in the study. The first five patients will have the Retroject device placed over their eye for 30 seconds and then removed. Assuming no issues, then it will be placed on the eye for one minute. The second group of patients (3 total) will have the Retroject device placed on the eye and then an injection of ethacrynic acid into the episcleral vein. The third group of patients (12 total) will have the Retroject device placed on the eye and then will be randomized in a 2:1 ratio to receive either an ethacrynic acid injection or a balanced salt solution injection. All 20 patients will then return for intraocular pressure measurements on days 1, 2, 3, and 7 as well as 6 weeks after injection. In addition, the patients will undergo pre and post intervention corneal endothelial assessments (endothelial cell count, shape analysis, and pachymetry). Potential safety issues are unlikely and include bleeding, infection, pain, ototoxicity, or temporary or permanent loss of vision.

ELIGIBILITY:
Inclusion Criteria:

* age 55 years or older of both sexes
* IOP >20 mmHg on maximal treatment
* <20/200 visual acuity
* willing to sign informed consent forms

Exclusion Criteria:

* monocular patients with bleeding disorders
* patients on anticoagulant or antiplatelet medications
* patients who had prior laser surgeries (SLT or ALT)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular pressures (IOP) lowering effect | Days 1, 2, 3, and 7, and 6 weeks after injection
  The patients will then return for intraocular pressure measurements on days 1, 2, 3, and 7 as well as 6 weeks after injection. Differences in baseline IOP versus post-injection IOP will be calculated for each patient.

OTHER OUTCOMES:
Corneal endothelial cell counts | 6 weeks after injection
  Pre and post injection (6 weeks) endothelial counts will be performed for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Rand Allingham, MD, Principal Investigator — Duke University Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States